CLINICAL TRIAL: NCT02829645
Title: Evaluation of the Clinical, Neuropsychological and Psychosocial Situation of Patient With Eating Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UF 8854
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Eating Disorders
Keywords: eating disoders; neuropsychology; pronostic
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eating disorders (Other)
  Interventions: Other: Clinical assessment

INTERVENTIONS:
Other: Clinical assessment — Clinical assessment with questionnaires

SUMMARY:
Eating disorders (ED) are serious mental illnesses with an excess mortality and many affects in the quality of life of patients and thier relatives. Management of ED is very difficult : the prognosis remains relatively poor both in terms of remission rate and quality of life. In this context, the contribution of new strategies for pathophysiological exploration and the development of therapeutic options are crucial.

In this project the investigators aim to constitute un cohort of patients from a day unit specialized in the management of ED. A prospective follow-up will be offered to patients to assess their clinical and psycho-social evolution. The overall objective is to identify which factors are prognostic of clinical improvement of the ED. We also want to better characterize patients that will migrate from diagnosis to another.

DETAILED DESCRIPTION:
The investigators propose to assess, with a cohort of patients with ED the prognostic value of cognitive abnormalities associated with ED (cognitive flexibility and central coherence) They will recruit 370 patients suffering from a current ED (anorexia, bulimia, binge eating disorder, Eating disorder not otherwise specified).

Each patient will be reassessed every year for 3 years.

ELIGIBILITY:
Inclusion criteria:

* respond to DSM 4 criteria for ED
* Age 15 to 65 years
* Signing an informed consent.
* Affiliated to a social security scheme or being the beneficiary of such a scheme.

Exclusion criteria:

* Manifest inability of the subject to understand / perform clinical and neuropsychological evaluations and tasks
* Major protected by law (guardianship)
* Privation of liberty by judicial or administrative decision
* Pregnant or lactating women

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of remission rates | At the inclusion and at 12, 24 and 36 months
  study of remission rates frequency at 12 months depending on the Brixton score assessed at baseline (assessment of cognitive flexibility). Remission is defined as disappearance of ED Diagnostic and Statistical Manual (DSM) criteria.

SECONDARY OUTCOMES:
score to another neuropsychological test (Iowa gambling task (IGT) | At the inclusion and at 12, 24 and 36 months
  Study of remission rates frequency at 12 months depending on the IGT score (decision making) assessed at baseline
scores to another other neuropsychological test : Rey-Osterrieth complex figure | At the inclusion and at 12, 24 and 36 months
  Study of remission rates frequency at 12 months depending on the Rey figure assessed at baseline
scores to another neuropsychological test : D2 test of attention | At the inclusion and at 12, 24 and 36 months
  Study of remission rates frequency at 12 months depending on the D2 test (attention) assessed at baseline

IPD SHARING:
Plan to Share IPD: No